CLINICAL TRIAL: NCT00480129
Title: The Anti-allergic Effects of Specific Probiotics - a Double Blind Clinical Study
Brief Title: The Anti-allergic Effects of Specific Probiotics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Ontario Ministry of Agriculture, Food and Rural Affairs (Other Government)
Responsible Party: Principal Investigator, Gregor Reid, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 12885
Record Dates: First submitted 2007-05-25; First posted 2007-05-30 (Estimated); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Allergic Rhinitis
Keywords: grass allergies,; ragweed allergies,; probiotics, lactobacillus,; bifidobacterium,; functional foods,; yogurt,; inflammatory cytokines
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Probiotics; Blood Specimen Collection; Nasal Lavage

INTERVENTIONS:
Behavioral: Probiotic or placebo yogurt consumed daily
Device: Mini Rhinoconjunctivitis Quality of Life Questionnaire
Procedure: Blood sample
Procedure: Nasal lavage

SUMMARY:
We hypothesize that specifically selected probiotics can alleviate symptoms of allergy in lactose tolerant individuals. Two strains of probiotics, Lactobacillus rhamnosus GR-1, and Bifidobacterium adolescentis 7007-05 will be used to create a yogurt product. Additionally a non-probiotic yogurt product will also be made as a placebo. Allergy sufferers will be asked to consume one of the two types of yogurts (blinded) for two months. During the two months there will be 3 sampling days, for blood samples and nasal lavage samples. Additionally Mini Rhinoconjunctivitis Quality of Life Questionnaires will be filled out weekly over the two months. After the two months of perceived responses as well sample analysis we should have a better idea of how these specific probiotic effect the immune system and allergies.

DETAILED DESCRIPTION:
Probiotics are "live microorganisms which when administered in adequate amounts confer a health benefit on the host". Many studies have been performed which indicate that probiotics can temporarily modify the composition of gut microbiota, and potentially these can reduce susceptibility to allergy (Noverr & Huffnagle, 2005) (Tannock et al. 2000), leading to health benefits for the host. Numerous studies show that these benefits include ones primed through the immune response of the host.

Animals maintained free of microorganisms have drastic abnormalities in their immune response. These germ-free animals have altered Peyer's Patches, reduced levels of IgA associated with increased risk for gastrointestinal infections, and they are unable to develop oral tolerance to ingested antigens (Moreau et al. 1988). When these animals are later colonized by normal intestinal bacteria, they overcome their past deficiencies, and have a restored ability for oral tolerance. This allows for the blockade of IgE production which is a key factor in allergic disease (Moreau et. al 1988).

Studies on inflammatory bowel disease patients have shown that certain probiotics can actually reduce inflammation and diminish disease (Bruzzese et al. 2004) (Baroja et al. submitted). The former study investigated 75 children, while our study (Baroja) showed down regulation of inflammation in 8/20 inflammatory bowel diseased patients. Allergic disease is almost non-existent in underdeveloped countries where, interestingly, fermented foods are consumed regularly. This differs considerably from the numerous allergies and lack of fermented food intake in the Western World. Investigators hypothesize that the human gut ecosystem has evolved to require daily intake of lactic acid bacteria (Molin 2001), and these bacteria maintain immunological regulation which protects against allergic sensitization and development of allergic disease.

Recent studies have shown that probiotics do have a significant influence on allergic reactions. The consumption of Lactobacillus rhamnosus GG by pregnant women lowered the occurrence of babies born with atopic dermatitis compared to those births from women who had not consumed the probiotic (Kalliomaki et al. 2001). Another study on 27 infants suffering from atopic eczema, showed that probiotic-supplemented formula decreased the severity of the condition (Isolauri et al 2000). The efficacy of probiotics in treating allergy has been further shown with Bifidobacterium longum BB536 in which it relieved Japanese cedar tree pollinosis, probably through the modulation of Th2-skewed immune response (Xiao et al. 2006). Another Japanese study showed that a synbiotic L. casei subsp. casei with dextran was an effective supplement for the prevention and treatment of allergic reactions cedar pollen (Ogawa et al. 2006). Not all studies have shown benefits, and one performed in teenagers and young adults allergic to birch pollen and apple food, showed no effect on intermittent symptoms of atopic allergy and/or mild asthma. We have now isolated strains of bifidobacteria from the stool of subjects with no history of any allergy, and these along with two lactobacilli probiotics have shown strong anti-allergy potential in vitro. In short, there is evidence to indicate that studies are worthwhile using food based probiotics, if not to completely prevent allergies, but to contribute towards their alleviation.

Objective 1. We will examine the cell types in nasal cavity with the expectation that this will shift as the probiotics are consumed, with a decrease in number of eosinophils, characteristic of late-phase allergic inflammatory symptoms, as the study progresses, and a corresponding decrease in neutrophils.

Objective 2. We will characterize the subject's sensitivities to inhalant seasonal and potentially year-round allergens. Routine RAST tests will be performed at the beginning of the study to test sensitivity towards mixed grasses, mixed trees, mixed weeds, mixed molds, ragweed, house dust, cat dander and dog dander. From this we will be able to differentiate subjects who are highly susceptible to allergy and those moderately susceptible. At the end of the trial we will perform further RAST tests using ragweed and mixed grass allergens, with the anticipation that the probiotic treatment with anti-allergic strains will decrease the subject's sensitivity to those particular allergens, while those receiving regular yogurt will have no effect.

Objective 3. We will identify changes in serum cytokine levels that would indicate a shift from an inflammatory state to one of reduced inflammation. We anticipate that the presence of inflammatory cytokines, IL-5, IL-4 and IL-13 will be decreased as the subject's intestinal flora is boosted by the anti-allergic probiotics; likewise, the presence of anti-inflammatory cytokines, IL-10, TGFβ2, IFN-γ will be increased by the treatment. This shift in cytokine production should be reflected in reduced allergic symptoms. In addition, Affymetrix Human Genome U133 Plus 2.0 Arrays will be performed on selected blood samples to characterize immunological signal transduction pathways activated by the probiotic bacteria.

Objective 4. We will characterize the perceived effects of anti-allergic strains of probiotics using a questionnaire. Subjects will self-administer validated Mini Rhinoconjunctivitis Quality of Life Questionnaire (MiniRQLQ)© (Juniper et al., 2000) on day 0 and weekly during the study period. The questionnaire includes 14 questions in five domains: activity limitations, practical problems and nose symptoms, eye symptoms and other symptoms. The questions are answered on scale 0-6 (from not troubled to extremely troubled) depending how troubled the subjects have been due to their nose/eye symptoms during the past week. Possible lung symptoms (cough, dyspnoea and wheezing) will be recorded separately using the same scale. This perceived effect may actually be the single most important outcome to our study. If the samples actually do show a decrease in inflammatory cytokines etc. but the subject does not perceive any changes to their allergy symptoms, then the probiotics cannot be stated to have affected the allergic response. We hope that all shifts in cytokine and cellular levels towards the anti-inflammatory state are reflected in the subject's awareness of decreased allergy symptoms.

At the end of this study we hope to know whether or not regular and probiotic yogurts have the potential to alleviate symptoms of allergic rhinitis, as well as down regulate the inflammatory processes in humans. It is anticipated that at least one of the yogurts will show promise in this regard. However, even a negative result would be informative, as the experiments will show us how consumers respond physiologically to different fermented food.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of allergic rhinitis based on sneeze attacks, runny/blocked/itchy nose in the absence of a common cold during the previous 12 months.
* History of positive skin prick test or blood radio-allergosorbent test (RAST) to grass and/or ragweed pollen

Exclusion Criteria:

* Ongoing allergen immunotherapy
* upper respiratory tract infection
* Pregnancy
* Clinical history of lactose-intolerance or allergies to cow-milk

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-05 (Actual); Primary Completion 2007-09 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Inflammatory versus anti-inflammatory serum cytokine fluctuations | 2 months
Allergen specific IgE fluctuations | 2 months
Type 2 T helper cell to Type 1 T helper cell ratios | 2 months
T regulatory cell production of interleukin-10 | 2 months
Cell count and type fluctuations in nasal lavage samples | 2 months
Protein concentration fluctuations in nasal lavage samples | 2 months

SECONDARY OUTCOMES:
Mini Rhinoconjunctivitis Quality of Life Questionnaire | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Gregor Reid, PhD, Principal Investigator — Lawson Health Research Institute - Canadian Research and Development Centre for Probiotics
Locations (1):
- Lawson Health Research Institute - Canadian Research and Development Centre for Probiotics, London, Ontario, Canada

REFERENCES:
- [Background] Molin G. Probiotics in foods not containing milk or milk constituents, with special reference to Lactobacillus plantarum 299v. Am J Clin Nutr. 2001 Feb;73(2 Suppl):380S-385S. doi: 10.1093/ajcn/73.2.380s. PMID 11157345
- [Background] Noverr MC, Huffnagle GB. The 'microflora hypothesis' of allergic diseases. Clin Exp Allergy. 2005 Dec;35(12):1511-20. doi: 10.1111/j.1365-2222.2005.02379.x. PMID 16393316
- [Result] Naclerio RM, Meier HL, Kagey-Sobotka A, Adkinson NF Jr, Meyers DA, Norman PS, Lichtenstein LM. Mediator release after nasal airway challenge with allergen. Am Rev Respir Dis. 1983 Oct;128(4):597-602. doi: 10.1164/arrd.1983.128.4.597. PMID 6354022
- [Result] Belda J, Parameswaran K, Keith PK, Hargreave FE. Repeatability and validity of cell and fluid-phase measurements in nasal fluid: a comparison of two methods of nasal lavage. Clin Exp Allergy. 2001 Jul;31(7):1111-5. doi: 10.1046/j.1365-2222.2001.01133.x. PMID 11468003
- [Result] Bruzzese E, Raia V, Gaudiello G, Polito G, Buccigrossi V, Formicola V, Guarino A. Intestinal inflammation is a frequent feature of cystic fibrosis and is reduced by probiotic administration. Aliment Pharmacol Ther. 2004 Oct 1;20(7):813-9. doi: 10.1111/j.1365-2036.2004.02174.x. PMID 15379842
- [Result] Isolauri E, Arvola T, Sutas Y, Moilanen E, Salminen S. Probiotics in the management of atopic eczema. Clin Exp Allergy. 2000 Nov;30(11):1604-10. doi: 10.1046/j.1365-2222.2000.00943.x. PMID 11069570
- [Result] Kalliomaki M, Salminen S, Arvilommi H, Kero P, Koskinen P, Isolauri E. Probiotics in primary prevention of atopic disease: a randomised placebo-controlled trial. Lancet. 2001 Apr 7;357(9262):1076-9. doi: 10.1016/S0140-6736(00)04259-8. PMID 11297958
- [Result] Moreau P, Paul P, Rouas-Freiss N, Kirszenbaum M, Dausset J, Carosella ED. Molecular and immunologic aspects of the nonclassical HLA class I antigen HLA-G: evidence for an important role in the maternal tolerance of the fetal allograft. Am J Reprod Immunol. 1998 Sep;40(3):136-44. doi: 10.1111/j.1600-0897.1998.tb00405.x. PMID 9764357
- [Result] Ogawa T, Hashikawa S, Asai Y, Sakamoto H, Yasuda K, Makimura Y. A new synbiotic, Lactobacillus casei subsp. casei together with dextran, reduces murine and human allergic reaction. FEMS Immunol Med Microbiol. 2006 Apr;46(3):400-9. doi: 10.1111/j.1574-695X.2006.00046.x. PMID 16553814
- [Result] Tannock GW, Munro K, Harmsen HJ, Welling GW, Smart J, Gopal PK. Analysis of the fecal microflora of human subjects consuming a probiotic product containing Lactobacillus rhamnosus DR20. Appl Environ Microbiol. 2000 Jun;66(6):2578-88. doi: 10.1128/AEM.66.6.2578-2588.2000. PMID 10831441
- [Result] Xiao JZ, Kondo S, Yanagisawa N, Takahashi N, Odamaki T, Iwabuchi N, Miyaji K, Iwatsuki K, Togashi H, Enomoto K, Enomoto T. Probiotics in the treatment of Japanese cedar pollinosis: a double-blind placebo-controlled trial. Clin Exp Allergy. 2006 Nov;36(11):1425-35. doi: 10.1111/j.1365-2222.2006.02575.x. PMID 17083353
- [Derived] Koyama T, Kirjavainen PV, Fisher C, Anukam K, Summers K, Hekmat S, Reid G. Development and pilot evaluation of a novel probiotic mixture for the management of seasonal allergic rhinitis. Can J Microbiol. 2010 Sep;56(9):730-8. doi: 10.1139/w10-061. PMID 20921983